CLINICAL TRIAL: NCT00647933
Title: An Open-label, Single Center Trial to Assess the Pharmacokinetics, Pharmacodynamics and Safety of Org 36286 After a Single Subcutaneous Dose in Healthy Female Volunteers Whose Pituitary Function is Suppressed by Lyndiol®.
Brief Title: An Open-label, Single Center Trial to Assess the Pharmacokinetics, Pharmacodynamics and Safety of Org 36286 (P07004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P07004; 38802
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Infertility
Keywords: Females; Corifollitropin alfa; Antibodies; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; Noracycline; Ethinyl Estradiol; Lynestrenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Org 36286 15 μg + Lyndiol® (Experimental): After a pill-free period of 7 days, participants took 1 oral tablet of Lyndiol® (50 μg ethinylestradiol + 2.5 mg lynestrenol) daily for a total period of at least 6 weeks to suppress endogenous gonadotropin secretion. After 3 weeks of Lyndiol® intake, participants received a single subcutaneous dose of Org 36286 15 μg.
  Interventions: Drug: Org 36286; Drug: Lyndiol®
- Org 36286 30 μg + Lyndiol® (Experimental): After a pill-free period of 7 days, participants took 1 oral tablet of Lyndiol® (50 μg ethinylestradiol + 2.5 mg lynestrenol) daily for a total period of at least 6 weeks to suppress endogenous gonadotropin secretion. After 3 weeks of Lyndiol® intake, participants received a single subcutaneous dose of Org 36286 30 μg.
  Interventions: Drug: Org 36286; Drug: Lyndiol®
- Org 36286 60 μg + Lyndiol® (Experimental): After a pill-free period of 7 days, participants took 1 oral tablet of Lyndiol® (50 μg ethinylestradiol + 2.5 mg lynestrenol) daily for a total period of at least 6 weeks to suppress endogenous gonadotropin secretion. After 3 weeks of Lyndiol® intake, participants received a single subcutaneous dose of Org 36286 60 μg.
  Interventions: Drug: Org 36286; Drug: Lyndiol®
- Org 36286 120 μg + Lyndiol® (Experimental): After a pill-free period of 7 days, participants took 1 oral tablet of Lyndiol® (50 μg ethinylestradiol + 2.5 mg lynestrenol) daily for a total period of at least 6 weeks to suppress endogenous gonadotropin secretion. After 3 weeks of Lyndiol® intake, participants received a single subcutaneous dose of Org 36286 120 μg.
  Interventions: Drug: Org 36286; Drug: Lyndiol®

INTERVENTIONS:
Drug: Org 36286 — Subcutaneous Org 36286
  Other Names: Corifollitropin alfa
Drug: Lyndiol® — Lyndiol® (50 μg ethinylestradiol + 2.5 mg lynestrenol) tablets orally once a day for 6 weeks.
  Other Names: 50 μg ethinylestradiol + 2.5 mg lynestrenol

SUMMARY:
The objectives of this study were to study the pharmacokinetics, pharmacodynamics and safety of Org 36286 after a single subcutaneous administration in healthy females.

ELIGIBILITY:
Inclusion Criteria:

* Good physical and mental health;
* Body Mass Index between 18 and 29 kg/m^2;
* Good venous accessibility;

Exclusion Criteria:

* Clinically relevant abnormal blood chemistry, hematology and/or urinalysis at screening;
* Hypertension (sitting diastolic blood pressure > 90 mmHg and/or systolic blood pressure > 150 mmHg);
* Contraindications for the use of oral contraceptives or gonadotropins;
* PAP-smear (= III) according to the Papanicolaou classification;
* History of endocrine abnormalities such as hyperprolactinaemia, polycystic ovary syndrome or any evidence of ovarian dysfunction;
* Primary ovarian failure;
* Ovarian cysts or enlarged ovaries, not related to polycystic ovarian disease;
* Any ovarian and/or abdominal abnormality that would interfere with adequate ultrasound investigation;
* Ovarian surgery;
* Smoking more than 10 cigarettes or equivalents a day;
* History (within 12 months) of alcohol or drugs abuse;
* Blood donation (> 200 ml) within 90 days prior to screening;
* Administration of investigational drugs within 90 days prior to start Org 36286.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2000-06; Primary Completion 2000-12 (Actual); Study Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Maximum number of follicles >= 5 mm (nmax) | Days 2 - 35
Mean dose-normalized maximum plasma concentration (Cmax) post single dose Org 36286 | Days 1 - 15
Mean dose-normalized area under the curve (AUC) post single dose Org 36286 | Days 1 - 15
Mean total plasma clearance (CL) post single dose Org 36286 | Days 1 - 15
Number of participants with an adverse event (AE) | Start of treatment up to day 28

SECONDARY OUTCOMES:
Day on which the number of follicles >= 5 mm was equal to nmax for the first time (dmax) | Days 2 - 35
Total number of follicles >= 5 mm per day | Days 2 - 35